CLINICAL TRIAL: NCT04693910
Title: Development and Evaluation of the Effectiveness of a Multimedia-based Hormonal Therapy Information Program for Patients With Prostate Cancer
Brief Title: Multimedia-based Hormonal Therapy Information Program for Patients With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hui Chien, RN PhD Associate Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201602024B0C501
Record Dates: First submitted 2020-12-23; First posted 2021-01-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Prostatic Neoplasms
Keywords: prostate cancer; hormonal therapy; multimedia; self-efficacy; positive thinking
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimedia information group (Experimental): The experimental group received a weekly multimedia hormone therapy information program for 6 weeks.
  Interventions: Other: Multimedia-Based Hormone Therapy Information Program
- Routine care group (No Intervention): The control group will receive routine care.

INTERVENTIONS:
Other: Multimedia-Based Hormone Therapy Information Program — The multimedia hormone therapy information program lasted 6 weeks and covered 6 topics, namely the recognition of hormone therapy and multimedia information programs, mindfulness, exercise, stress relief, positive thinking, and prevention or reduction of fatigue.
  Arms: Multimedia information group

SUMMARY:
This study takes place in the Divisions of Urology. Patients who have only received hormonal therapy will be enrolled. Patients will be randomly sorted into an experimental group and a control group after completing a pretest questionnaire. The experimental group will receive the the multimedia hormone therapy information program once per week for 6 consecutive weeks, while the control group will receive routine care. The follow-up data collections will be completed at 8 and 12 weeks after the pretest. For quantitative measurement, the main variables will be social support, self-efficacy, quality of life, and positive thinking.

DETAILED DESCRIPTION:
This study takes place in the Divisions of Urology at Chang Gung Memorial Hospitals. Patients who have only received hormonal therapy will be enrolled. With reference to past research findings, self-efficacy theory, and experts' advice, a multimedia hormone therapy information program was developed. The multimedia hormone therapy information program covered 6 topics, namely the recognition of hormone therapy and multimedia information programs, mindfulness, exercise, stress relief, positive thinking, and prevention or reduction of fatigue. A pilot study will be conducted to check the feasibility of intervention study design and the effectiveness of the program will be tested. Patients will be randomly sorted into an experimental group (multimedia information group, n = 36 to 40) and a control group (routine care group, n = 36 to 40) after completing a pretest questionnaire. The experimental group will receive the multimedia information intervention once per week for 6 consecutive weeks, while the control group will receive routine care. The follow-up data collections will be completed at 8 and 12 weeks after the pretest. For quantitative measurement, the main variables will be social support, self-efficacy, quality of life, positive thinking, and satisfaction with program. Generalized Estimating Equations (GEEs) will be used to o analyze data.

ELIGIBILITY:
Inclusion Criteria:

1. patients with prostate cancer who were receiving hormonal therapy
2. patients were at least 20 years old
3. patients were ability to communicate in Chinese or Taiwanese
4. the married partner agrees to study together, or the single patient has a cohabitation partner who agrees to study together.
5. patients or family have a smart phone or tablet and can connect to the Internet.

Exclusion Criteria:

1. having a history of other cancers
2. unknown diagnosis of prostate cancer or unknown disease status
3. patients who received chemotherapy, radiotherapy, radical prostatectomy or other treatments for prostate cancer in the past
4. having history of mental disorder, e.g., phobia, obsessive-compulsive disorder, generalized anxiety, , major depression, mania, manic-depressive psychosis, or dementia
5. the score of Eastern Cooperative Oncology Group performance is ≧ 2

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | pretest
  A total of 39 items, including five subdimensions, namely, physical well-being, social/family well-being, emotional well-being, functional well-being, and prostate cancer subscales. A 5-point scoring method was adopted. Higher scores indicate higher quality of life
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 8 weeks after the pretest
  A total of 39 items, including five subdimensions, namely, physical well-being, social/family well-being, emotional well-being, functional well-being, and prostate cancer subscales. A 5-point scoring method was adopted. Higher scores indicate higher quality of life
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | 12 weeks after the pretest
  A total of 39 items, including five subdimensions, namely, physical well-being, social/family well-being, emotional well-being, functional well-being, and prostate cancer subscales. A 5-point scoring method was adopted. Higher scores indicate higher quality of life
The Positive Thinking Scale | pretest
  A total of 18 items, including two subscales of personal satisfaction and goal pursuit. A five-point (1-5) scoring method was used. Higher scores indicate a higher level of positive thinking
The Positive Thinking Scale | 8 weeks after the pretest
  A total of 18 items, including two subscales of personal satisfaction and goal pursuit. A five-point (1-5) scoring method was used. Higher scores indicate a higher level of positive thinking
The Positive Thinking Scale | 12 weeks after the pretest
  A total of 18 items, including two subscales of personal satisfaction and goal pursuit. A five-point (1-5) scoring method was used. Higher scores indicate a higher level of positive thinking
The Hormonal Dimension of The Expanded Prostate Cancer Index Composite | pretest
  11 items were used, the score of each item ranges from 0 to 100 points. Higher scores indicate fewer hormonal symptoms.
The Hormonal Dimension of The Expanded Prostate Cancer Index Composite | 8 weeks after the pretest
  11 items were used, the score of each item ranges from 0 to 100 points. Higher scores indicate fewer hormonal symptoms.
The Hormonal Dimension of The Expanded Prostate Cancer Index Composite | 12 weeks after the pretest
  11 items were used, the score of each item ranges from 0 to 100 points. Higher scores indicate fewer hormonal symptoms.

SECONDARY OUTCOMES:
The General Self-Efficacy Scale | pretest
  The total scale contains 10 items and a 4-point (1-4) scoring method was adopted. Higher scores indicate higher self-efficacy
The General Self-Efficacy Scale | 8 weeks after the pretest
  The total scale contains 10 items and a 4-point (1-4) scoring method was adopted. Higher scores indicate higher self-efficacy
The General Self-Efficacy Scale | 12 weeks after the pretest
  The total scale contains 10 items and a 4-point (1-4) scoring method was adopted. Higher scores indicate higher self-efficacy
The Social Support Scale | pretest
  A total of 16 items, including four sub-scales of emotional, informational, appraisal, and instrumental support. A 4-point scoring method (0-3) was used. Higher scores indicate stronger support.
The Social Support Scale | 8 weeks after the pretest
  A total of 16 items, including four sub-scales of emotional, informational, appraisal, and instrumental support. A 4-point scoring method (0-3) was used. Higher scores indicate stronger support.
The Social Support Scale | 12 weeks after the pretest
  A total of 16 items, including four sub-scales of emotional, informational, appraisal, and instrumental support. A 4-point scoring method (0-3) was used. Higher scores indicate stronger support.

OTHER OUTCOMES:
Basic and disease information list 1 | pretest
  Age
Basic and disease information list 2 | pretest
  Education level
Basic and disease information list 3 | pretest
  Marital status
Basic and disease information list 4 | pretest
  Religion
Basic and disease information list 5 | pretest
  Occupation
Basic and disease information list 6 | pretest
  Annual family income (NTD)
Basic and disease information list 7 | pretest
  Number of children
Basic and disease information list 8 | pretest
  Join a support group
Basic and disease information list 9 | pretest
  Time since diagnosis (months)
Basic and disease information list 10 | pretest
  Tumor-node-metastasis Cancer stage
Basic and disease information list 11 | pretest
  Gleason score
Basic and disease information list 12 | pretest
  Treatment
Basic and disease information list 13 | pretest
  History of chronic disease
Basic and disease information list 14 | pretest
  Living status
Basic and disease information list 15 | pretest
  Height in centimetre
Basic and disease information list 16 | pretest
  Body Mass Index in kg/m2 will be computed from height and body weight
Basic and disease information list 17 | pretest
  Body weight in kilograms
Basic and disease information list 18 | pretest
  Waist circumference in centimetre
Basic and disease information list 19 | pretest
  Serum Prostatic Specific Antigen level
Basic and disease information list 20 | 8 weeks after the pretest
  Serum Prostatic Specific Antigen level
Basic and disease information list 21 | 12 weeks after the pretest
  Serum Prostatic Specific Antigen level
Basic and disease information list 22 | pretest
  Perceived health status. A 11-point (0-100) scoring method was used. Higher scores indicate better health condition.
Basic and disease information list 23 | 8 weeks after the pretest
  Perceived health status. A 11-point (0-100) scoring method was used. Higher scores indicate better health condition.
Basic and disease information list 24 | 12 weeks after the pretest
  Perceived health status. A 11-point (0-100) scoring method was used. Higher scores indicate better health condition.
List of satisfaction with Program | 8 weeks after the pretest
  Five items were self-designed to understand the satisfaction of men in the experimental group. A 11-point (0-100) scoring method was used. Higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hui Chien, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences, Taipei city, Taiwan
Locations (1):
- Chang Gung Memorial Hospital at Linkou, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data of this study will be kept and managed by PI of Ching-Hui Chien.

REFERENCES:
- [Background] Cary KC, Singla N, Cowan JE, Carroll PR, Cooperberg MR. Impact of androgen deprivation therapy on mental and emotional well-being in men with prostate cancer: analysis from the CaPSURE registry. J Urol. 2014 Apr;191(4):964-70. doi: 10.1016/j.juro.2013.10.098. Epub 2013 Oct 29. PMID 24184370
- [Background] Cella DF, Tulsky DS, Gray G, Sarafian B, Linn E, Bonomi A, Silberman M, Yellen SB, Winicour P, Brannon J, et al. The Functional Assessment of Cancer Therapy scale: development and validation of the general measure. J Clin Oncol. 1993 Mar;11(3):570-9. doi: 10.1200/JCO.1993.11.3.570. PMID 8445433
- [Background] Cheung SK, Sun SY. Assessment of optimistic self-beliefs: further validation of the Chinese version of the General Self-Efficacy Scale. Psychol Rep. 1999 Dec;85(3 Pt 2):1221-4. doi: 10.2466/pr0.1999.85.3f.1221. PMID 10710976
- [Background] Chien CH, Liu KL, Chien HT, Liu HE. The effects of psychosocial strategies on anxiety and depression of patients diagnosed with prostate cancer: a systematic review. Int J Nurs Stud. 2014 Jan;51(1):28-38. doi: 10.1016/j.ijnurstu.2012.12.019. Epub 2013 Feb 8. PMID 23398917
- [Background] Chien CH, Chuang CK, Liu KL, Wu CT, Pang ST, Tsay PK, Chang YH, Huang XY, Liu HE. Effects of individual and partner factors on anxiety and depression in Taiwanese prostate cancer patients: A longitudinal study. Eur J Cancer Care (Engl). 2018 Mar;27(2):e12753. doi: 10.1111/ecc.12753. Epub 2017 Sep 18. PMID 28921733
- [Background] Cockle-Hearne J, Barnett D, Hicks J, Simpson M, White I, Faithfull S. A Web-Based Intervention to Reduce Distress After Prostate Cancer Treatment: Development and Feasibility of the Getting Down to Coping Program in Two Different Clinical Settings. JMIR Cancer. 2018 Apr 30;4(1):e8. doi: 10.2196/cancer.8918. PMID 29712628
- [Background] Diefenbach MA, Mohamed NE, Butz BP, Bar-Chama N, Stock R, Cesaretti J, Hassan W, Samadi D, Hall SJ. Acceptability and preliminary feasibility of an internet/CD-ROM-based education and decision program for early-stage prostate cancer patients: randomized pilot study. J Med Internet Res. 2012 Jan 13;14(1):e6. doi: 10.2196/jmir.1891. PMID 22246148
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Esper P, Mo F, Chodak G, Sinner M, Cella D, Pienta KJ. Measuring quality of life in men with prostate cancer using the functional assessment of cancer therapy-prostate instrument. Urology. 1997 Dec;50(6):920-8. doi: 10.1016/S0090-4295(97)00459-7. PMID 9426724
- [Background] Keating NL, O'Malley A, Freedland SJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy: observational study of veterans with prostate cancer. J Natl Cancer Inst. 2012 Oct 3;104(19):1518-23. doi: 10.1093/jnci/djs376. No abstract available. PMID 23210129
- [Background] Chien CH, Chuang CK, Liu KL, Wu CT, Pang ST, Chang YH. Health-Related Quality of Life and Its Associated Factors in Prostate Cancer Patients Who Receive Androgen Deprivation Therapy. Cancer Nurs. 2021 Jan/Feb;44(1):E34-E42. doi: 10.1097/NCC.0000000000000752. PMID 31743152
- [Background] Chien CH, Chuang CK, Liu KL, Pang ST, Wu CT, Chang YH. Exploring the Positive Thinking of Patients With Prostate Cancer: Self-efficacy as a Mediator. Cancer Nurs. 2022 Mar-Apr 01;45(2):E329-E337. doi: 10.1097/NCC.0000000000000868. PMID 32649333
- [Background] Loiselle CG, Edgar L, Batist G, Lu J, Lauzier S. The impact of a multimedia informational intervention on psychosocial adjustment among individuals with newly diagnosed breast or prostate cancer: a feasibility study. Patient Educ Couns. 2010 Jul;80(1):48-55. doi: 10.1016/j.pec.2009.09.026. Epub 2009 Oct 24. PMID 19854604
- [Background] Van Gerven PW, Paas F, Van Merrienboer JJ, Hendriks M, Schmidt HG. The efficiency of multimedia learning into old age. Br J Educ Psychol. 2003 Dec;73(Pt 4):489-505. doi: 10.1348/000709903322591208. PMID 14713374
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Wootten AC, Abbott JA, Meyer D, Chisholm K, Austin DW, Klein B, McCabe M, Murphy DG, Costello AJ. Preliminary results of a randomised controlled trial of an online psychological intervention to reduce distress in men treated for localised prostate cancer. Eur Urol. 2015 Sep;68(3):471-9. doi: 10.1016/j.eururo.2014.10.024. Epub 2014 Oct 28. PMID 25454611
- [Background] Zhang Q, Zhao H, Zheng Y. Effectiveness of mindfulness-based stress reduction (MBSR) on symptom variables and health-related quality of life in breast cancer patients-a systematic review and meta-analysis. Support Care Cancer. 2019 Mar;27(3):771-781. doi: 10.1007/s00520-018-4570-x. Epub 2018 Nov 28. PMID 30488223
- [Derived] Chien CH, Liu KL, Chuang CK, Wu CT, Chang YH, Yu KJ. Multimedia-based hormone therapy information program for patients with prostate cancer: the result of a randomized pilot study. Sci Rep. 2023 Dec 27;13(1):23022. doi: 10.1038/s41598-023-50006-6. PMID 38155164